CLINICAL TRIAL: NCT00590772
Title: Phase 4- The Role of Montelukast on Perennial Rhinitis and Associated Sleep Disturbance and Daytime Somnolence
Brief Title: The Role of Montelukast in Rhinitis and Sleep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Timothy Craig, Principal Investigator, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 2003-114; Merck Grant #IISP ID# 20030
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Perennial Allergic Rhinitis
Keywords: sleep; somnolence; allergies; rhinitis; fatigue
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Sleepiness; Hypersensitivity; Rhinitis; Fatigue | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- montelukast (Active Comparator): montelukast 10 mg daily
  Interventions: Drug: montelukast
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: montelukast — 10 mg po each day (compared to placebo for 2 weeks)
  Other Names: Singulair
  Arms: montelukast
Drug: placebo — placebo for 2 weeks
  Arms: Placebo

SUMMARY:
The hypothesis is that a leukotriene receptor antagonist (LRA), montelukast, will decrease nasal congestion leading to increased patency of the nose and a decrease in nighttime sleep fragmentation in individuals with year round allergic rhinitis or perennial allergic rhinitis (PAR). This decrease in sleep fragmentation will reduce daytime somnolence and fatigue.

DETAILED DESCRIPTION:
Montelukast is a once daily LRA indicated for the treatment of allergic rhinitis and asthma, which is both safe and effective. Documented improvement in nasal congestion has been showed in patients with both seasonal and perennial allergic rhinitis. As demonstrated in recent publications, we fully anticipate that nasal congestion will be reduced in individuals afflicted with AR treated with montelukast. We have previously documented that a decrease in nasal congestion is associated with improved subjective sleep quality and subjective improvement in daytime somnolence. However, we have not demonstrated a cause and effect relationship. Currently, we have a study being performed that will allow us to assess the effect of nasal steroids on objective sleep by collecting data using a traditional overnight sleep test in subjects with congestion. We have not yet determined if subjective instruments for daytime somnolence correlate with objective measurements of improved daytime sleepiness. The purpose of this protocol will be three fold. First, we hope to determine the effectiveness of montelukast to reduce fatigue, somnolence and improve sleep, by reducing nasal congestion in allergic rhinitis. Two, we will assess the statistical relation between subjective instruments for sleepiness. Lastly, we want to determine the most appropriate test to use to determine daytime sleepiness or somnolence in patients with seasonal allergen induced congestion and daytime sleepiness.

We will be dosing montelukast once a day, which is the manufacturer's suggested dosing schedule. Active drug will be compared to a placebo vehicle, which will mimic the active drug. With the proposed design study, a run-in period is not essential; however, to establish baseline symptoms and adherence to therapy, we have chosen a 1-week run-in while on placebo. After run-in, patients will be randomized to either active drug or placebo after baseline questionnaires and other data are collected. A daily diary to determine symptoms of allergic rhinitis and nighttime disturbance, as well as, daytime fatigue will be issued and expected to be completed daily. Two weeks after randomization, a follow-up will be scheduled in order to insure compliance, to collect diaries, administer questionnaires, and start the second treatment phase. After this visit study subjects will enter a 1-week wash-out and have a return visit before being randomized to the alternative arm. At six weeks, subjects will again be seen to insure compliance and administer questionnaires. The study will conclude following six-weeks. The data used for analyses will be the data collected during the last week of each randomized period. This will decrease cross over affect, typically seen in classical cross over studies, since there will be only a short washout between cross over.

Subjects selected for this study will have a history of allergic rhinitis and a positive RAST or skin test to a perennial (year round) allergen and have symptoms that correlate with this allergen. If prior skin test or RAST is not available, a skin test will be performed to confirm allergic rhinitis. The patients will be seen in either the Allergy, Asthma, and Respiratory research center or the GCRC. All care and all studies will be done free of charge at no cost to the subject. Each subject will be compensated for his or her participation as outlined below.

Patients will also be expected to have fatigue, daytime somnolence and poor sleep on study entry. An instrument to access the degree of fatigue, sleepiness and sleep quality will not only be required to be positive, but also must designate the symptom as greater than 50% on a severity rating.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will include:

1. Age 16 to 65.
2. History of allergic rhinitis.
3. The ability to be placed on placebo without significant compromise in the quality of life.
4. General good health.
5. Ability to comply with the protocol and sign an informed consent.
6. Have daytime sleepiness by history.
7. Have poor sleep by history.
8. Have fatigue by history.
9. Have a skin test or RAST test to a perennial allergen (indoor mold, dog, cat, mite) with correlating symptoms.

Exclusion Criteria:

1. Age fewer than 16 or over 65 years.
2. A history of sleep apnea.
3. Atopic diseases other than allergic rhinitis, such as atopic dermatitis or asthma.
4. Non-allergic rhinitis.
5. Obesity.
6. Inability to tolerate montelukast.
7. Significant other diseases as determined by the investigator.
8. Use of a research medication within 30 days.
9. Use of a nasal steroid or topical antihistamine or decongestant within 30 days.
10. Use of beta-blockers, antidepressants, oral decongestants, oral steroids, or H2-blockers.
11. Excessive use of alcohol or drug abuse.
12. Inability to stop medication use during run-in period.
13. Use of an oral antihistamine within 1 week of enrollment.
14. Failed to have benefit when montelukast was used for rhinitis or asthma in the past

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

REFERENCES:
- [Result] Santos CB, Hanks C, McCann J, Lehman EB, Pratt E, Craig TJ. The role of montelukast on perennial allergic rhinitis and associated sleep disturbances and daytime somnolence. Allergy Asthma Proc. 2008 Mar-Apr;29(2):140-5. doi: 10.2500/aap.2008.29.3097. PMID 18430310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients screened in research laboratory
Pre-assignment Details: Patients had a run-in to determine symptoms and only if they had congestion with poor sleep and daytime somnolence were they enrolled
Groups:
- Group 1: subjects were randomized to placebo or active drug and then cross over to opposite; however, the details of the randomization are no longer available.
Period: Overall Study
Arm/Group | Group 1
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: cross over
Arm/Group | Group 1
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — data are not available at this time
  Male | NA — data are not available at this time
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fatigue and Daytime Sleepiness at 2 Weeks
Description: Daytime sleepiness was assessed on a scale of 0 (none) to 4 with 4 being severe.
  To determine improvement of daytime sleepiness with active therapy we used a scale of 0 to 4 with 0 being no improvement and 4 being maximal improvement.
  To determine improvement of daytime fatigue with active therapy we used a scale of 0 to 4 with 0 being no improvement and 4 being significant improvement.
  For all three above we used data from the last 3 days were averaged and mean of change for each day.
Time Frame: baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 31 | 31
units on a scale
  daytime sleepiness | -0.64 (NA) — data are no longer available | 0.13 (NA) — data are no longer available
  improved daytime sleepiness | 0.46 (NA) — data are no longer available | -0.25 (NA) — data are no longer available
  improved daytime fatigue | 0.43 (NA) — data are no longer available | -0.32 (NA) — data are no longer available

ADVERSE EVENTS:
Arm/Group | Montelukast | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No